CLINICAL TRIAL: NCT02413125
Title: Comparison of Nasal Saline Irrigation Bottle Contamination Between Two Solutions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Stephen Bakos, MD, Resident Physician, University of Virginia
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17882
Record Dates: First submitted 2015-02-18; First posted 2015-04-09 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Sinusitis
MeSH Terms: conditions — Sinusitis | interventions — Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ChitoRino irrigation solution (Experimental): The study participants will be provided a NeilMed irrigation bottle and instructed to administer 1 packet of ChitoRhino irrigation solution (premixed from manufacturer containing sea salt, Chitosan, and sodium bicarbonate). An informational sheet regarding care and cleaning of the irrigation bottle will be provided during the initial visit. Participants will be instructed to complete up to three nasal saline irrigations daily for 1 month and keep a log to determine compliance. After 1 month of use, the irrigation bottle will be returned at a second study visit.
  Interventions: Device: ChitoRhino irrigation solution
- Normal saline solution (Experimental): The study participants will be provided a NeilMed irrigation bottle and instructed to administer nasal saline (250mL of 0.9% sodium chloride) irrigation solution. An informational sheet regarding care and cleaning of the irrigation bottle will be provided during the initial visit. Participants will be instructed to complete up to three nasal saline irrigations daily for 1 month and keep a log to determine compliance. After 1 month of use, the irrigation bottle will be returned at a second study visit.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Device: ChitoRhino irrigation solution — ChitoRhino irrigation solution has been developed with chitosan, a natural polysaccharide demonstrated to have antibacterial and antifungal properties. This polysaccharide has beneficial properties in multiple clinic applications including wound healing and post-operative sinus surgery. Chitosan's antimicrobial function develops from its polycationic structure. Chitosan interacts with the negatively charge bacterial wall, leading to disruption and cell lysis.
  Arms: ChitoRino irrigation solution
Drug: Normal saline — Most nasal irrigations use normal saline (0.9% sodium chloride), which approximates the physiological concentration of plasma in the blood. The saline solution is used to flush the nose of mucous and allergens.
  Arms: Normal saline solution

SUMMARY:
Rhinosinusitis is one of the most prevalent diseases within the United States and leads to decreased quality of life for patients suffering from this condition. A foundation in treatment for rhinosinusitis is nasal saline irrigations, which are administered through an irrigation bottle. The irrigation bottles are prone to contamination by bacterial and fungal species despite proper maintenance.

A new commercially available irrigation solution has been created using chitosan, a natural polysaccharide with antibacterial and antifungal properties. This research project will examine the ability of chitosan to decrease or prevent contamination of irrigation bottles after 1 month use by adult patients with rhinosinusitis.

Participants in this project will use either saline or chitosan irrigation solution for 1 month and then switch to the other solution for 1 month. Following 1 month of use, the irrigation bottles will be cultured to determine if chitosan irrigation solution decreased the contamination of the irrigation bottles.

DETAILED DESCRIPTION:
Rhinosinusitis is one of the most prevalent diseases in the United States with an estimated 31 million adults diagnosed with this condition. The annual health care burden has been estimated to exceed 5.8 billion dollars. Unfortunately, the underlying etiology of rhinosinusitis is not fully understood and may encompass multiple factors including: anatomic variations, impaired immune function, ciliary dysfunction, seasonal allergies, aspirin allergy, and bacterial biofilms. There are a wide variety of treatment options aimed at reducing the symptoms of rhinosinusitis with nasal saline irrigations (NSI) being one of the foundations for therapeutic intervention.

The benefits of NSI in rhinosinusitis in reducing nasal symptoms have been demonstrated in multiple reports. The mechanisms in which NSI exerts its beneficial effects are not fully understood, though multiple theories exist including: improvement in mucociliary function, decreased nasal mucosal edema, and removal of infectious debris and allergens. NSI are administered intranasally with the use of an irrigation bottle with a wide variety of brands commercially available for patients to select. In the Department of Otolaryngology-Head and Neck Surgery Clinic at the University of Virginia Health System, NeiMed bottles are provided to patients who are diagnosed with rhinosinusitis. In addition, the patients are given an informational sheet regarding the care and cleaning of these irrigation bottles. Unfortunately, irrigation bottles can become colonized with bacteria including: Staphylococcus aureus, Streptococcus pneumonia, Pseudomonas aeruginosa, and Candida species. The contamination of irrigation bottles can be a nidus for continued bacterial introduction into the nasal cavity and therefore decreasing the beneficial effects of NSI.

Recently, a novel commercially available irrigation solution, the ChitoRhino, has been developed with chitosan, a natural polysaccharide demonstrated to have antibacterial and antifungal properties. This polysaccharide has beneficial properties in multiple clinic applications including wound healing and post-operative sinus surgery. Chitosan's antimicrobial function develops from its polycationic structure. Chitosan interacts with the negatively charge bacterial wall, leading to disruption and cell lysis. There is a paucity of literature examining the beneficial effect of chitosan in decreasing bacterial contamination in irrigation bottles. This project represents a pilot study investigating the antimicrobial effects of chitosan in irrigation bottles for patients with rhinosinusitis.

ELIGIBILITY:
Inclusion Criteria:

* participants will be: 18 years old or older,
* diagnosed with rhinosinusitis based on history and physical examination performed for clinical care
* intervention to be prescribed would include nasal irrigation,
* able to understand and comply with the study protocol instructions, including the return the irrigation bottles

Exclusion Criteria:

* children less than 18 years old,
* unable to understand or perform the saline irrigations, or protocol instructions including the return the irrigations bottles after 1 month of use
* prisoners
* those with shellfish allergies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-02; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Bacterial contamination of nasal saline irrigation bottle following normal saline solution assessed by performing a bacterial culture | 1 month
  Patients will be provided an irrigation bottle and instructed to use normal saline for 1 month. Following this period, the saline irrigation bottle will be collected and a bacterial culture of the irrigation bottle will be performed to determine the bacterial contamination present following use.
Bacterial contamination of nasal saline irrigation bottle following ChitoRhino irrigation solution assessed by performing a bacterial culture | 1 month
  Patients will be provided an irrigation bottle and instructed to use the ChitoRhino irrigation solution for 1 month. Following this period, the saline irrigation bottle will be collected and a bacterial culture of the irrigation bottle will be performed to determine the bacterial contamination present following use.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen R Bakos, M.D./Ph.D., Principal Investigator — Department of Otolaryngology-Head and Neck Surgery University of Virginia Health System
Locations (1):
- Department of Otolaryngology-Head and Neck Surgery at the University of Virginia Health System, Charlottesville, Virginia, United States